CLINICAL TRIAL: NCT00934791
Title: Single Center, Open-label Randomized Prospective Trial: Effect of Sirolimus on Polycystic Liver Disease
Brief Title: Polycystic Liver Disease in Kidney Transplant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to inadequate enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Principal Investigator, Patrick G. Dean, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-004315
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Polycystic Liver Disease
Keywords: Kidney Transplant; Autosomal dominant polycystic kidney disease; Polycystic liver disease
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant | interventions — Tacrolimus; Sirolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Tacrolimus, mycophenolate mofetil, and prednisone
  Interventions: Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Drug: Prednisone
- Sirolimus Group (Active Comparator): Sirolimus, mycophenolate mofetil, and prednisone
  Interventions: Drug: Sirolimus; Drug: Mycophenolate Mofetil; Drug: Prednisone

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus 6-10 mg/day (maintain trough levels of 8-10 ng/mL)
  Other Names: Prograf
  Arms: Control Group
Drug: Sirolimus — Sirolimus 3-5 mg/day (maintain high-performance liquid chromatography (HPLC) blood level 10-15 ng/mL)
  Other Names: Rapamune; Rapamycin
  Arms: Sirolimus Group
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 750 mg twice daily
  Other Names: Cellcept
Drug: Prednisone — Prednisone tapered to 5 mg/day by day 92
  Other Names: Deltasone

SUMMARY:
The purpose of this study is to see if one kind of immunosuppressive drug has better effects for the patient's polycystic liver disease than another type. Tacrolimus and Sirolimus are the two immunosuppressive drugs that will be compared for this study. Both drugs have been commonly prescribed to prevent rejection.

DETAILED DESCRIPTION:
Autosomal dominant polycystic kidney disease (ADPKD) is a life-threatening monogenic disease with a prevalence of 1 in 400-1000 livebirths. ADPKD is caused by mutations to polycystic kidney disease 1 gene (PKD1) (approximately 85% of cases) or polycystic kidney disease 2 gene (PKD2) (the remaining 15%) gene, encoding polycystin-1 (PC1) and polycystin-2 (PC2), respectively. PC1 is a putative cell-surface, receptor-like protein with yet to-be-identified ligand(s), and PC2 a channel protein with a high conductance to Ca2+.

Polycystic liver disease (PLD) is the most common extra-renal manifestation in ADPKD, present in > 90% of ADPKD patients by age 30. Liver cysts in ADPKD originate from biliary micro-hamartoma or focal proliferations of biliary ductules and from peribiliary glands. Excessive proliferation of biliary epithelial cells, combined with neovascularization, altered cell-extracellular matrix (ECM) interaction/ECM remodeling and cAMP-mediated fluid secretion, is required for the development and expansion of PLD liver cysts.

PLD may become symptomatic with acute complications such as cyst hemorrhage, rupture and infection. Chronic symptoms are frequently associated with massively enlarged PLD, including abdominal distension and pain; dyspnea; gastroesophageal reflux and early satiety which may lead to malnutrition; mechanical lower back pain; obstruction of the inferior vena cava, hepatic and portal veins (leading to dialysis-associated hypotension, hepatic venous outflow obstruction, and portal hypertension) and biliary obstruction. Currently, apart from invasive interventions such as cyst aspiration with sclerosis, cyst fenestration combined hepatic resection and cyst fenestration, liver transplantation and, rarely, selective hepatic artery embolization, no medical therapy is available.

The objective of this study is to conduct a prospective, open-label, randomized trial to examine the effect of sirolimus on total liver volume in kidney transplant recipients with ADPKD.

Four weeks following kidney transplant, subjects will undergo iothalamate clearance measurement, 24-hour urine collection and protein measurement and physical examination by a transplant surgeon. Patients will be randomized to receive either sirolimus-based immunosuppression or to continue tacrolimus-based immunosuppression unless one of the following conditions are noted:

1. Complications of the kidney transplant incision, including, but not limited to: superficial wound infection, deep wound infection, and fascial dehiscence
2. Iothalamate clearance measurement less than 40 mL/min/1.72m^2
3. Urinary protein excretion greater than 800 mg/24 hours. Subjects with the above conditions will continue to receive tacrolimus-based immunosuppression at the discretion of the treating physician/surgeon.

Enrolled subjects will undergo abdominal and pelvic CT scans within 3 months before or after kidney transplantation and at one, two, and three years after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years old) with stage IV or V chronic kidney due to ADPKD
* Primary kidney transplant
* Living or deceased donor kidney transplant
* Estimate total liver volume of 2.5 to 7.5 L
* In addition, at the discretion of the principal investigator(s), certain subjects with numerous liver cysts but with liver volume < 2.5 liters may be enrolled.

Exclusion Criteria:

* Pediatric patients (< 18 years of age)
* Patients with Body Mass Index (BMI) greater than or equal to 40 kg/m^2
* Multi-organ transplant (kidney-liver, etc.)
* When people who have one blood type receive blood from someone with a different blood type, it may cause their immune system to react. This is called (ABO) incompatibility. ABO-incompatible or positive cross-match recipients
* Patients with severe hyperlipidemia (serum cholesterol > 350 mg/dl or serum triglycerides > 500 mg/dl)
* Patients with leukopenia (WBC < 3000 10/ml)
* Patients unwilling to return to the transplant center for late follow-up visits
* Patients who are currently pregnant or breast-feeding or who expect to be pregnant during the study period
* Female patients of child bearing potential and men with sexual partners of child bearing potential who do not agree to use a medically accepted method of contraception during the study period
* Patients who are not eligible for Thymoglobulin induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Dean, M.D., Principal Investigator — Mayo Clinic; QI Qian, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants were enrolled in the study in Rochester, Minnesota. One participant withdrew before doing any part of the study; he was not randomized to a group.
Period: Overall Study
Arm/Group | Control Group | Sirolimus Group
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Sirolimus Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Liver Volume at 2 Years After Kidney Transplantation
Description: Liver volume at 2 years will be compared between the sirolimus and control (tacrolimus) groups using analysis of covariance (ANCOVA).
Time Frame: 2 years
Population: This study was terminated due to inadequate enrollment, no data was collected on the participant.
Arm/Group | Control Group | Sirolimus Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group | Sirolimus Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated due to inadequate enrollment, no data was collected on the participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No